CLINICAL TRIAL: NCT05458713
Title: The Effect of Laser Acupuncture in Different Meridians on the Autonomic Nervous System and Its Brain Mechanisms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, Taiwan (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Tu Cheng-Hao, Associate Professor, China Medical University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MOST 111-2320-B-039-031-MY2
Record Dates: First submitted 2022-07-10; First posted 2022-07-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Laser Acupuncture; Meridian; Heart Rate Variability; Brain Mechanism
Keywords: pericardium meridian; laser acupuncture; pulse rate variability; Resting-state functional magnetic resonance imaging; bladder meridian

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PC6 High Energy group (Experimental): The participants of this group will be irradiated with a 4mm probe for 60 seconds with an output power of 100mW on PC6 (acupoint Neiguan).
  Interventions: Device: Laser acupuncture
- PC6 Low Energy group (Experimental): The participants of this group will be irradiated with a 4mm probe for 20 seconds with an output power of 100mW on PC6 (acupoint Neiguan).
  Interventions: Device: Laser acupuncture
- PC6 Placebo group (Placebo Comparator): The participants of this group will be irradiated with a 4mm probe for 0 seconds with an output power of 100mW on PC6 (acupoint Neiguan).
  Interventions: Device: Laser acupuncture
- BL65 High Energy group (Active Comparator): The participants of this group will be irradiated with a 4mm probe for 60 seconds with an output power of 100mW on BL65 (acupoint Shugu).
  Interventions: Device: Laser acupuncture
- BL65 Low Energy group (Active Comparator): The participants of this group will be irradiated with a 4mm probe for 20 seconds with an output power of 100mW on BL65 (acupoint Shugu).
  Interventions: Device: Laser acupuncture
- BL65 Sham group (Sham Comparator): The participants of this group will be irradiated with a 4mm probe for 0 seconds with an output power of 100mW on BL65 (acupoint Shugu).
  Interventions: Device: Laser acupuncture

INTERVENTIONS:
Device: Laser acupuncture — Irradiate acupoints with low power laser

SUMMARY:
Traditional Chinese acupuncture has a history of several thousand years. The World Health Organization has published guidelines describing the efficacy of acupuncture in the cure or relief of 64 different symptoms and conditions as one of the most representative intangible cultural heritage of humanity. In recent years, the applications of laser acupuncture, or so-called low-level laser therapy which are belong to the domain of photobiomodulation therapy, become widespread. Laser acupuncture is not only applicate to stimuli specific areas in need, but also one of non-invasive intervention technic with hurtles intervention, no hematoma, bleeding or swelling unpleasant feeling after intervention, which could be more accepted by children, weakness people, and patients who afraid of acupuncture. However, the underlined mechanisms and the neural pathway of laser acupuncture are still obscure.

The inconsistent results from previous studies have been reported that laser acupuncture stimulation on the Neiguan (PC 6), the acupoint of Pericardium meridian, could affect the autonomic nerve system in terms of heart rate, blood pressure, activities of sympathetic and/or parasympathetic nerves. The results of previous studies on the changes of autonomic nervous system (ANS) caused by laser acupuncture on Neiguan (PC6), an acupoint of the pericardium meridian, have been inconsistent. Our preliminary results show that laser acupuncture on PC6 seems to have a biphasic dosage effect on the ANS changes. However, little is known about the possible central mechanisms underpinned these ANS changes. In addition, whether laser acupuncture on different meridians will also induce a biphasic dosage effect on the ANS is still unknown. Therefore, the main purposes of this project are: 1) to explore the changes of ANS and associated brain networks by applying laser acupuncture with on PC6 different intensities; and 2) to explore whether applying laser acupuncture on different meridians will have different ANS and related brain network responses. In this two-year, single-blind, parallel experiment design project, the recruited healthy subjects will randomly assign to the group with high energy density, low energy density, or no energy of laser acupuncture on PC6 (in first year) or on Shugu (in second year), which is an acupoint of the bladder meridian (BL65). Via a non-invasive wearable photoplethysmography, the peripheral pulse rate variability will be calculated as the index of ANS changes. In addition, the resting-state functional MRI scans will be performed before and after laser acupuncture to explore the immediate changes in the brain networks that may regulates the activity of ANS. The investigators hope that through the application of modern scientific methods to probe the meridian phenomenon in Chinese medicine, The investigators can further understand the neurological mechanisms of the meridian and provide a new insight for the traditional meridian theory of Chinese medicine.

DETAILED DESCRIPTION:
Acupuncture therapy is an important branch of traditional Chinese medicine for the treatment of clinical diseases. However, due to its more invasive treatment, some patients (such as children or patients with trauma to acupoints) are not suitable for this treatment. In recent years, laser acupuncture (irradiating acupoints with low-power lasers) has gradually become popular in the clinical application of traditional Chinese medicine because of its non-invasiveness, no pain, and few side effects. There are many domestic and foreign case reports showing that it may have curative effects . For example, in patients with severe peripheral facial nerve palsy who have not been significantly improved for 12 years, after four months of laser acupuncture intervention, the affected side of the eye can be completely closed, and the sagging facial muscles on the affected side can be significantly raised. For severe sciatica patients with an average Visual Analogue Scale (VAS) score of 9.6, the pain was relieved by more than half after the first laser acupuncture, and their symptoms disappeared completely after the 56th intervention. For children with low acceptance of traditional acupuncture, some studies have also pointed out that laser acupuncture treatment for about 12 times a month can effectively improve children with tension-type cerebral palsy due to central regulation problems. of muscle spasm, especially in the biceps brachii, iliopsoas, thigh adductor muscle group, etc., the effect is more significant. For carpal tunnel syndrome, studies have also confirmed that after about 20 laser acupuncture interventions a month, the symptoms of peripheral carpal tunnel syndrome have been significantly improved.

Although the above-mentioned clinical cases and studies have shown that laser acupuncture may have clinical efficacy in some diseases, its mechanism is not yet clear. At present, most of its clinical efficacy is explained by the mechanism of photomodulation therapy, that is, after laser stimulation, it will change the redox reaction of local mitochondria, promote the synthesis of ATP and increase the body's energy source, and can activate endocrine regulation, regulate the concentration of neurotransmitters, anti-inflammatory, and restore blood circulation, thereby resulting in a series of clinical effects such as repair and functional recovery. However, laser acupuncture has not accumulated as many research results as traditional acupuncture, and the mechanism through which the central nervous system achieves clinical efficacy has not been extensively explored, let alone its relationship with the meridians. Several pilot studies have previously performed laser acupuncture at different acupoints and observed changes in heart rate variability (HRV) to explore whether laser acupuncture could alter the autonomic nervous system. However, due to the differences in operating parameters such as wavelength, time, output power, probe size, and even energy density of laser acupuncture, the research results on whether laser acupuncture affects HRV and even the autonomic nervous system are inconsistent. Some reports show that laser acupuncture at Neiguan can increase the overall power of HRV, but other studies show no significant change. If the effect of laser acupuncture on sympathetic or parasympathetic nerve activity is further analyzed, it has been reported that in subjects on night shifts, laser acupuncture at Neiguan acupoint can significantly increase parasympathetic nerve activity and reduce sympathetic nerve activity . However, in patients with chronic insomnia, laser acupuncture at Neiguan acupoint significantly increased sympathetic nerve activity and decreased parasympathetic nerve activity. Therefore, there is still a lot of room to be clarified and explored in the way of laser acupuncture at Neiguan, the influence on the autonomic nervous system, and its possible central nervous system.

Research Objectives Past research on light modulation therapy has pointed out that its dose effect often presents a biphasic dosage effect, that is, the Arndt-Schulz law: after the dose exceeds the minimum threshold, the effect of the low dose area increases with the dose increase, but The effect in high-dose regions decreases with increasing dose. Therefore, the inconsistent results of laser acupuncture at Neiguan acupoint on HRV and even the autonomic nervous system may also be related to the biphasic dose effect. The purpose of this study is to 1) explore the changes in the autonomic nervous system and brain activities caused by laser acupuncture of different intensities on Neiguan point; 2) to explore whether laser acupuncture is accompanied by different autonomic nerve responses and brain activities on acupoints of different meridians. In this study, the investigators expected to recruit healthy subjects, and in a parallel experimental design, the three-intensity laser was applied to the Neiguan point on the pericardium meridian or the Shugu point (BL65) of the bladder meridian with high, low and no intensities Acupuncture, through PRV changes (such as heartbeat, systolic blood pressure, diastolic blood pressure, heartbeat interval, low frequency power, high frequency power, low/high frequency power ratio, etc.), observe the effect on the autonomic nervous system. In addition, resting-state fMRI was also used to understand the corresponding changes in the regulation of autonomic nervous system-related brain network activity before and after laser acupuncture. Through these designs, the investigators hope to explore the relationship between laser acupuncture dose, autonomic changes, and changes in related brain network activity to clarify their possible neural mechanisms. And by extension, compare it with the bladder meridian of Foot Taiyang, analyze the meridian phenomenon contained in the pericardium meridian of handicapped Jueyin, and conduct a pilot study on its possible clinical treatment of neural mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between the ages of 20 and 55.
2. Body Mass Index (BMI) should fall between 18.5 and 24 kg/m2.
3. Voluntarily sign the subject's consent form reviewed and approved by the human trial committee, indicating voluntary participation in the research.

Exclusion Criteria:

1. Those diagnosed with chronic diseases such as coronary artery disease, diabetes, hypertension, hyperlipidemia, cancer, etc.
2. With the brain diseases, such as epilepsy, stroke, Parkinson's disease, dementia, brain tumor, traumatic brain injury, head trauma or brain surgery, etc.
3. The positive result for wrist Tinel sign, or who have experienced neurological symptoms such as median nerve compression recently and during the experiment.
4. Patients with mental disorders, such as major depression, bipolar disorder, generalized anxiety disorder, claustrophobia, schizophrenia, etc.
5. Cannot follow the instructions to perform the experiment due to hyperactivity and agitation.
6. Taken neuropsychiatric drugs (such as sleeping pills, anti-anxiety drugs) or pain relievers and other drugs that affect nerve activity in the past three months.
7. Pregnant, plan to pregnant, or menopausal women.
8. Having metal implants in the body, or equipping with a pacemaker.
9. With scars or open wounds at the acupoints selection site, or the skin condition at the site may affect the selection of acupoints or laser acupuncture.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-13 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity in brain | 500 seconds before and 30 seconds after laser acupuncture intervention
  The changes of functional connectivity with laser acupuncture intervention

SECONDARY OUTCOMES:
Heart rate variability (HRV) | 500 seconds before and 30 seconds after laser acupuncture intervention
  The changes of heart rate variability (HRV) with laser acupuncture intervention

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No